CLINICAL TRIAL: NCT00962182
Title: Effect of a Cocktail of Two Common Enzyme Supplements on Celiac Disease Patients With Persistent Seropositivity
Brief Title: Study of Enzyme Supplements to Treat Celiac Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Heim Pal Children's Hospital (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Ilma R Korponay-Szabo, Professor, Heim Pal Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-03
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Celiac Disease; Dermatitis Herpetiformis
Keywords: celiac disease; transglutaminase antibody
MeSH Terms: conditions — Celiac Disease; Dermatitis Herpetiformis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Enzyme treatment (Experimental): Enzyme for 12 weeks
  Interventions: Drug: STAN1
- Placebo control (Placebo Comparator): Placebo enzyme for 12 weeks
  Interventions: Drug: Placebo enzyme
- Enzyme + gluten (Experimental): Enzyme and 500 mg gluten b.i.d. for 12 weeks
  Interventions: Drug: STAN1+gluten

INTERVENTIONS:
Drug: STAN1 — 3-4 capsules/day at meals
  Arms: Enzyme treatment
Drug: Placebo enzyme — 3-4 capsules/day at meals
  Arms: Placebo control
Drug: STAN1+gluten — 3-4 capsules/day at meals plus 500 mg gluten b.i.d
  Arms: Enzyme + gluten

SUMMARY:
The purpose of this study is to examine whether a cocktail of two common food-grade enzyme supplements leads to decrease of serum activity markers in celiac disease patients insufficiently treated by previous gluten exclusion.

DETAILED DESCRIPTION:
Celiac disease is genetically determined abnormal immune response to gluten, a component of wheat, rye and barley proteins that cause damage to the villous structure in the small bowel. The active disease is characterized by the induction of gluten-dependent autoantibodies to transglutaminase type-2, which are sensitive and specific non-invasive markers of gluten-sensitivity. Gluten-free diet normally leads to clearance of antibodies from serum in 6-12 months. Persistent seropositivity is a problem in patients who only incompletely exclude gluten or frequently transgress the diet. In such cases, damage of the small bowel may persist and complications may occur at higher frequency. The central hypothesis to be tested is that enzyme treatment designed to degrade a certain amount of gluten before absorption in the gastrointestinal tract will lead to a clinically meaningful decrease in auto-antibody levels in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Celiac disease diagnosed by small intestinal biopsy
* More than 12 months elapsed since initial diagnosis and start of the dietary treatment
* Evidence for ongoing active disease as verified by seropositivity or dermatitis herpetiformis rash
* Subject agrees to follow a gluten-free diet

Exclusion Criteria:

* Other gastrointestinal or hepatic disease besides celiac disease
* Selective IgA deficiency
* Use of dapsone or diaphenylsulfone
* Pregnancy and breast-feeding

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-08; Primary Completion 2014-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Negative seroconversion or a drop of more than 50% in anti-transglutaminase antibody blood levels by ELISA | 12 weeks

SECONDARY OUTCOMES:
Negative seroconversion or drop of at least two dilution steps in the EMA test | 12 weeks
Negative conversion for celiac antibodies in the blood by the rapid test | 12 weeks
Change in symptoms or rash (if any) | 12 weeks
Favorable changes in morphometry in small bowel biopsy specimens | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ilma Korponay-Szabo, M.D., Ph.D., Study Director — Heim Pal Children's Hospital
Locations (2):
- Hungary (2):
  - Heim Pal Children's Hospital, Budapest
  - University of Debrecen, Debrecen